CLINICAL TRIAL: NCT04160377
Title: A Clinical Trial of Fluvoxamine for Melancholia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lingjiang Li (Other)
Responsible Party: Sponsor-Investigator, Lingjiang Li, President of Chinese Psychiatry Society of Chinese Medical, Central South University
Organization: Central South University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-08-01-XY-0001
Record Dates: First submitted 2019-11-08; First posted 2019-11-13 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Depressive Disorder; Endogenous Depression; Melancholia
MeSH Terms: conditions — Depressive Disorder | interventions — Fluvoxamine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- melancholic depression (Experimental): patients with melancholic depression undergo the treatment of Fluvoxamine
  Interventions: Drug: Fluvoxamine
- non-melancholic depression (Experimental): patients with non-melancholic depression undergo the treatment of Fluvoxamine
  Interventions: Drug: Fluvoxamine

INTERVENTIONS:
Drug: Fluvoxamine — Fluvoxamine was assigned to be the treatment for the depression patients with melancholic features or not .
  Other Names: Fluvoxamine Maleate Tablets

SUMMARY:
This study aims at investigating the special effectiveness of antidepressant effect of Fluvoxamine for endogenous depression. The investigators also aim to assess the effect of Fluvoxamine on the multimodal magnetic resonance imaging(MRI), blood cytokines, feces bacteria flora and neuropsychological performance in depression patients with melancholic features. The investigators further aim to identify the predictors of Fluvoxamine's antidepressant effeect using the above techniques.

DETAILED DESCRIPTION:
This study aims at investigating the special effectiveness of antidepressant effect of Fluvoxamine for melancholia. The investigators also aim to assess the effect of Fluvoxamine on the multimodal magnetic resonance imaging(MRI), blood cytokines, feces bacteria flora and neuropsychological performance in depression patients with melancholic features. The investigators further aim to identify the predictors of Fluvoxamine's antidepressant effeect using the above techniques.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18-55 years, both sexes), with DSM-4 criteria for MDD without psychosis, as determined by a structured clinical interview Mini International Neuropsychiatric Interview
* Moderate to severe depression, as defined by a pretreatment score ≥17 on the HDRS-17 scale
* Informed consent to participate in this study
* ethinic Han, right-handed, Junior high school education or above

Exclusion Criteria:

* A history of bipolar disorder, schizophrenia, schizoaffective disorder, obsessive-compulsive disorder, panic disorder, or documented Axis II diagnoses; active suicidal intention, as determined by clinical interview
* Active or recent (<12 months) substance abuse or dependence; excluding nicotine
* Presence of ECT treatment in recent 6 months
* period of pregnancy or lactation
* hearing disorder or colour blindness
* Immediate relatives have bipolar disorder or mania disorder

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Hamilton Depression Rating Scale-17 item (HAMD-17) | Baseline, 2weeks, 1 months, 2 months
  Interview-based questionnaire used to measure the severity of depression. Consists of 17 items with a score calculated. Higher scores are associated with more severe depression.
Change in Hamilton Anxiety Rating Scale-14 item (HAMA-14) | Baseline, 1 months, 2 months
  Interview-based questionnaire used to measure the severity of anxiety. Consists of 14 items with a score calculated. Higher scores are associated with more severe anxiety.
Change in voxel-based morphometry of grey matter, white matter as assessed by structural magnetic resonancce imaging | Baseline, 2 months
  Participants will receive resting-state functional magnetic resonance imaging (MRI). Scans will be performed on a 3.0- T Siemens Magnetom Skyra scanner (Siemens Healthineers, Erlangen, Germany). During scanning, all participants were instructed to remain motionless, and to think of nothing in particular but to not fall asleep.
Change in Functional connectivity | Baseline, 2 months
  Change in Functional connectivity of the brain networks as assessed by measure of connectivity in multimodal MRI.

SECONDARY OUTCOMES:
Change in peripheral blood cytokines | Baseline, 1 months, 2 months
  Peripheral blood sample will be collected and the concentration of IL-6, TNF-α, and CRP will be assessed.
Change in feces bacterial flora | Baseline, 1 months, 2 months
  The objective of investigator is to characterize gut microbiome in patients with TRD. To explore the specific diversity of gut microbiome. The stool samples were collected in the collection kits at the baseline, and were frozen at -80 °C. After the process of DNA Purification, 16S rRNA Gene Amplification and Illumina MiSeq sequencing, the study finally find the abundance and diversity of microbiota.
Change in Congruent STROOP Time to Complete (Executive Function) | Baseline, 1 months, 2 months
  Stroop Colour Naming Test (STROOP) is a cognitive test designed to assess the ability to inhibit a prepotent response to reading words while performing a task that requires attention control. It comprises two sheets with 50 words on each, and each word is the name of a colour. On the first sheet, the Congruent STROOP Sheet, the word and ink colour match; on the Incongruent STROOP Sheet, the word and ink colour do not match. For each sheet, the patient has 4 minutes to name the ink colour of each word. When the patient finishes the sheet, or once 4 minutes is up, the clinician notes the time taken and counts the number of correct and incorrect responses. The scale ranges from 0-100, the higher score the greater the cognitive flexibility.
Change in DSST (Number of Correct Symbols) | Baseline, 1 months, 2 months
  Digit Symbol Substitution Test (DSST) is a cognitive test designed to assess psychomotor speed of performance requiring visual perception, spatial decision-making, and motor skills. It consists of 133 digits and requires the patient to substitute each digit with a simple symbol in a 90-second period. Each correct symbol is counted, and the total score ranges from 0 (less than normal functioning) to 133 (greater than normal functioning)." as a description of DSST.
Improvement on Snaith-Hamilton Pleasure Scale (SHAPS) | Baseline, 1 months, 2 months
  The Snaith-Hamilton Pleasure Scale (SHAPS) assesses the anhedonia symptoms of MDD patients, with higher score indicating more severe anhedonia. Evaluating the patient's pleasure experience and choosing the degree of agreement with the happy response in some pleasant situations, and each item was rated on a 4-point scale."1 = Strongly agree, 2 = agree, 3 = disagree and 4
  = strongly disagree" This scale evaluates the status of patients in the recent period of time, The total score of the scale is the sum of the scores of 14 items, with a total score of 14-56. The higher the total score, the more serious the anhedonia.
Young Manic Rating Scale (YMSR) | Baseline, 1 months, 2 months
  The YMSR assesses the manic symptoms of the subjects.
Life Event Scale (LES) | Baseline, 1 months, 2 months
  The LES assesses the effects of some life events on the subjects.
Beck Scale for Suicide Ideation（BSI） | Baseline, 1 months, 2 months
  The BSI assesses the Suicide Ideation of the subjects, including two time points, the latest week and when the subjects were the most depressive.
Hopkins Vocabulary Learning Test-Revised (HVLT-R) | Baseline, 1 months, 2 months
  The HVLT-R assesses the memory and the cognition of the subjects.
Sydney Melancholia Prototype Index (SMPI) | Baseline, 1 months, 2 months
  The SMPI aims to identify the melancholic and non-melancholic depression.
Generalized Anxiety Disoder-7 (GAD-7) | Baseline, 1 months, 2 months
  The GAD-7 aims to assesses the severity of anxious symtoms.
Self-reported Quick Inventory of Depressive Symptomatology (QIDS-SR) Scale | Baseline, 1 months, 2 months
  The QIDS-SR assesses the depressive symtoms in latest week of subjects quickly.
Dimensional Anhedonia Rating Scale (DARS) | Baseline, 1 months, 2 months
  The DARS assesses different dimensions in Anhedonia of the subjects.
Child Trauma Scale (CTQ) | Baseline, 1 months, 2 months
  The CTQ assesses child trauma happen to the subjects.
Sheehan Disability Scale (SDS) | Baseline, 1 months, 2 months
  The SDS assesses the impairment in the occupational, familial and social ability of the subjects.
Pittsburgh Sleep Quality Index (PSQI) | Baseline, 1 months, 2 months
  The PSQI assesses the sleep quality of the subjects.
Perceived Deficit Questionnaire for Depression (PDQ-D) | Baseline, 1 months, 2 months
  The PDQ-D assesses the perceived deficit of the subjects
Medication Adherence Rating Scale (MARS) | 1 months, 2 months
  The MARS assesses the medication adherence condition of the subjects
Rating Scale for Side Effects (SERS) | 1 months, 2 months
  The SERS assesses the side effects of medication condition in the subjects

OTHER OUTCOMES:
Halstead-Reitan neuropsychological test battery for adults（HRB） | Baseline, 1 months, 2 months
  Halstead-Reitan neuropsychological test battery for adults assesses the basic functions of the brain，including perception, orientation, attention, action speed and memory.
Wechsler Scale (Digital Span) | Baseline, 1 months, 2 months
  Wechsler Scale (Digital Span) assesses the Attention and short-term memory of the subjects.
Electroencephalogram (EEG) | Baseline, 2 weeks
  EEG Microstate Parameters data like"ECG QT Interval" or "EEG power in the alpha band, etc., were collected at a 5000 Hz sampling rate, using a 64-channel Ag-Cl electrode (Brain Products) for both resting-state and task-state.

CONTACTS AND LOCATIONS:
Overall Officials: Lingjiang Li, MD, Principal Investigator — Mental Health Institute, the Second Xiangya Hospital of Central South University
Locations (1):
- Mental Health Institute & Faculty of Psychiatry of The Second Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li X, Yan D, Liao M, Zhang L, Li Z, Liu B, Chen Y, Zhang Y, Liu J, Li L. Effect of fluvoxamine on plasma interleukin-6 in patients with major depressive disorder: a prospective follow-up study. Front Psychiatry. 2023 May 25;14:1163754. doi: 10.3389/fpsyt.2023.1163754. eCollection 2023. PMID 37304432